CLINICAL TRIAL: NCT02838394
Title: Does Site-specific Trigger Point Dry Needling Evoke Segmental Neuromodulation in the Lower Extremity and if so, do These Changes Make an Impact on the Subject's Disability?
Brief Title: Dry Needling and Functional Improvement
Acronym: DN
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: no clinician who will collect data
Sponsor: Brigham Young University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16225
Record Dates: First submitted 2016-07-18; First posted 2016-07-20 (Estimated); Last update posted 2024-04-25 (Actual); Status verified 2023-07

CONDITIONS: Myofascial Trigger Point Pain; Myofascial Pain Syndrome
MeSH Terms: conditions — Myofascial Pain Syndromes | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dry Needling (Experimental): Trigger points found in the gluteal region of one side (e.g. right) will be dry needled; presence of muscle twitching (which would signify appropriate needle insertion) will be documented.
  Interventions: Procedure: Dry needling
- Sham Dry Needling (Sham Comparator): Trigger points found in the gluteal region of one side (e.g. right) will be SHAM dry needled with blunted needles, no actual penetration through the skin will occur.
  Interventions: Other: Sham dry needling

INTERVENTIONS:
Procedure: Dry needling — Acupuncture filiform needles are inserted into myofascial trigger points
  Other Names: Trigger point dry needling, intramuscular needling
  Arms: Dry Needling
Other: Sham dry needling — Blunted needles will be pressed against the skin, but no actual penetration will occur
  Arms: Sham Dry Needling

SUMMARY:
Dry Needling (DN) is a skilled intervention that uses acupuncture filiform needles that are inserted into myofascial trigger points or other tissues underneath the skin. It is used to treat myofascial or neuromusculoskeletal pain and to improve movement impairments. Although more and more physical therapists add this treatment tool to their skill box, there is uncertainty about its working mechanism and its efficacy. The latter is partially due to the challenging task of finding and using a true control or sham treatment. The investigators will use blunted needles, which will not perforate the skin, as sham treatment.

This study will assess if DN of a trigger point in the gluteal muscles increases pain pressure threshold in that muscle, in another muscle innervated by the same segment (L4/5) and in an area not supplied by the same segment (i.e. the ipsilateral posterior shoulder). In addition, this study will assess if functionality, as measured by the Oswestry Disability Index (ODI) and 15-point Global Rating of Change Scale (GRoC) questionnaires, improves after 2-3 treatments (1 week) of DN.

DETAILED DESCRIPTION:
Background Dry Needling (DN) is a skilled intervention that uses acupuncture filiform needles that are inserted into myofascial trigger points or other tissues underneath the skin [Dunning]. Trigger points are spots in taut muscle fibers that can produce local and radiating pain when irritated, for example when pressed upon. Several theories on the etiology of trigger points exist, such as a local energy crisis and increased acetylcholine release due to mechanical muscle overuse [Bron]. The existence of trigger points is widely accepted [Hong], although there are also some vocal opponents [Quintner 2015, Quintner 1994].

The aim of DN is to treat myofascial or neuromusculoskeletal pain and improve movement impairments. The mechanism which with DN purportedly works has been the subject of debate for many years. It is generally accepted that the needle has to be inserted into a trigger point, where it will produce a local muscle twitch response and consequently 'inactivate' the trigger point [Dunning]. Some propose that the quick muscle contraction induces normalization of tissue pH and reduction of biochemical and neurotransmitters that stimulate pain receptors - a local response [Shah]. Others suggest that DN interrupts the trigger point's ongoing nociceptive input into the dorsal horn - a segmental response [Fernandez-de-las-Penas]. Others again submit that, because some trigger points affect limbic and dorsal hippocampus activity, DN might have a central response [Niddam].

The efficacy of DN is also not completely clear, but shows a trend. One early literature review and meta-analysis concluded that DN was not significantly superior to placebo control in regards to pain decrease [Tough]. However, since then several systematic reviews with meta-analyses [Tekin, Kietrys, Boyles] determined that the evidence suggested that DN for trigger point-derived pain was likely to be the most effective approach, was superior in decreasing pain compared to stretching and percutaneous electric nerve stimulation and at least as effective as manual trigger point release and other needling treatments. One literature analysis supports the use of DN not only for its immediate, but also short-term effectiveness in reducing pain in patients with upper quarter myofascial pain syndrome [Kietrys].

Controlled trials that assess DN efficacy either use 1) sham or control (such as no or an inactive treatment) or 2) other treatments (such as lidocaine injections, non-local DN, or "usual care", such as stretching and exercise) for the comparison group. A blunted needle that does not penetrate the skin is a good sham treatment [Streitberger] and has been recommended as adequate control. As discussed elsewhere [Streitberger], every needle penetration, be it at a trigger point or not, will induce physiological responses and are as such not appropriate to use as control.

Srbely et al. found that one intervention of trigger point stimulation with DN evoked palliative effects in other areas innervated by the same spinal segment. They dry needled trigger points in the supraspinatus and assessed pressure sensitivity changes in the infraspinatus (same segment, C5) and gluteus maximus (different segment, L4/5, S1). Their results suggest that pain pressure threshold was increased after 3 and 5 minutes of DN in the areas supplied by the C5 segment, but not in the area supplied by L4/5, S1.

The above named study only assessed immediate pain-related changes due to the intervention and did not assess functional improvements. The investigators of this study were not able to find any articles investigating this phenomenon in the lower extremity. This project will use a similar set up as the above study, but the subjects will receive sham DN, not real DN in a non-trigger point tissue (which, as explained above, will still elicit physiological effects and could have some segmental influence) as in the above named study. In addition, the investigators will explore if there are functional improvements in subjects receiving DN. Consequently, the investigators propose to perform the following controlled study that explores the questions 'Does site specific trigger point dry needling evoke segmental neuromodulation in the lower extremity and if so, do these changes make an impact on the subject's disability?'.

The aims are:

I) Regarding Pain

1. Assess if pain pressure threshold (PPT) decreases in the muscle that received DN
2. Assess if PPT decreases in the muscle that received sham DN (not perforating the skin)
3. Assess if low back pain decreases more in the treatment group compared to sham group

II) Regarding Functionality

1. Assess if the level of disability due to pain will be lower after one week of treatment in the subjects who received DN
2. Assess if the level of disability due to pain will be significantly lower in subjects who received DN compared to those who received sham

III) Regarding Mechanism

1. Assess if specific trigger point DN evokes segmental neuromodulation in the lower extremity; meaning that if a trigger point in a muscle that is innervated by a certain segment is DN, other trigger points in the same segment will exhibit decreased PPT as well.
2. Assess if PPT associated with trigger points in the infraspinatus change after DN the lower back

Our hypotheses are:

I)

* H1: PPT decreases in the gluteus maximus/medius after one week of DN
* H2: Trigger points that receive DN with sham needles (not perforating the skin) will not exhibit the same amount of decreased PPT compared to the trigger points that are DN with actual treatment DN

II)

* H3: Low back pain will decrease more in the treatment group compared to sham
* H4: The level of disability due to pain will decrease after one week of DN treatment
* H5: The level of disability due to pain will be significantly lower in subjects who received DN treatment compared to the subjects who received sham treatment

III)

* H6: Specific trigger point dry needling will evoke segmental neuromodulation in the lower extremity; meaning that if the investigators DN a trigger point in the gluteus maximus/medius, that are innervated by L4/L5, other trigger points in the same segment (i.e. multifidus at segment L4/5) will exhibit decreased PPT as well
* H7: PPT associated with trigger points in the infraspinatus will not change after DN the lower back Subjects will have been referred to Peaks Performance Physical Therapy (Baton Rouge, Louisiana) for diagnosis of 'trigger point gluteal muscles', 'myofascial pain', 'neuromuscular pain' or 'low back pain' (or similar) who demonstrate painful taut bands of tight muscle tissue in the gluteal muscles and infraspinatus and complain of radiating pain when point pressure is exerted onto that tight muscle tissue.

Methods

Prospective subjects will undergo physical examination by the co-author PC to identify inclusion and exclusion criteria.

The main inclusion criterion will be the presence of a painful trigger point in the gluteals (gluteus maximus or medius) and infraspinatus on the same side. The painful trigger point is defined as a distinct hypersensitive taut band within a muscle that begins to radiate diffuse pain into adjacent areas with sustained pressure. In keeping with the study conducted by Srbely et al. the investigators will only include trigger points with a baseline (pre-intervention) pain pressure threshold (PPT) value of 35 N or less in order to improve reliability of their detection. The precise location of each trigger point will be marked on the skin using a non-toxic marker for ease of follow-up identification.

If the patient is deemed eligible for the study, the investigating PT will explain the study to the prospective subject and he/she will be asked if he/she wants to participate. The PT will explain that the subject might not get the actual DN technique, but instead a sham. If the subject declines he/she will receive treatment as 'normal'. If he/she agrees, he/she will receive the informed consent to read and sign. If there are study-related questions they will be answered. After this the subject will fill out an intake sheet for demographic information, the modified Oswestry Disability Questionnaire (mOSW) [Copay] as well as a pain map and visual analog scale (VAS) for low back pain. The subject will then determine his/her group allocation by drawing a piece of paper out of an opaque envelope. This envelope will contain 40 pieces of paper; 20 of them will specify 'dry needling A' (for treatment), 20 will specify 'dry needling B' (for sham).

The rest of the physical therapy treatment will be pragmatic; the subject will receive mobilizations (no grade 5: high velocity low amplitude), exercises as indicated and DN for one week (2-3 visits). Grade 5 mobilizations (or manipulations) will be excluded as treatment option because they are believed to elicit neurophysiological effects, similar to DN, and might skew the results.

Study flow/ data intake

1. The investigators will measure pressure sensitivity via algometer in the gluteal muscles, the ipsilateral multifidus at level L4/5 and the ipsilateral infraspinatus.
2. The investigators will dry needle trigger points found in the gluteal region of one side (e.g. right) and document of muscle twitching (which would signify appropriate needle insertion) OR sham dry needle (with blunted needle, no actual penetration through the skin will occur)
3. Exercises will be performed as needed (pragmatic, but no manipulations). This regimen will be followed for maximally one week, (less, if pain is abolished).
4. At the end of the week PPT will be measured, VAS, the mOSW and the 15-point Global rating of change scales (GRoC) [Kamper] questionnaires will be given and results will be documented.

Data Analysis

PPT readings will be normalized to baseline scores so the focus is on the percent changes, not on the absolute changes in values.

* H1: baseline PPT measurements in the gluteus maximus/medius from 20 subjects who receive DN will be compared to post PPT measurements, taken after one week of DN will be analyzed using a paired t-test
* H2: change in PPT in the gluteus maximus/medius from 20 subjects who received DN will be compared to the change in PPT from 20 subjects who received sham DN will be analyzed with a 2-sample t-test
* H3: VAS score changes from 20 subjects who received DN will be compared to the VAS score changes from 20 subjects who received sham DN will be analyzed with a 2-sample t-test
* H4: The baseline mOSW scores from 20 subjects who received DN will be compared to the post treatment scores of the mOSW and will be analyzed with a paired t-test
* H5: The changes in mOSW and GRoC scale scores from 20 subjects who received DN will be compared to the changes in mOSW and GRoC scale scores from 20 subjects who received sham DN will each be analyzed with a 2-sample t-test
* H6: Pre- to post treatment changes in PPT in the gluteus maximus/medius will be compared to the changes measured in the multifidus at segment L4/5 and analyzed with a paired t-test
* H7: Pre- to post treatment changes in PPT in the gluteus maximus/medius will be compared to the changes measured in the infraspinatus and analyzed with a paired t-test

All significance levels will be set at 0.05. The minimally clinically important difference (MCID) for the VAS is 2 points [Childs], for the OSW it is 12.8 points [Copay] and the 'important improvement' for the GRoC is 5 points [Kamper].

ELIGIBILITY:
Inclusion Criteria:

* presence of at least one painful trigger point in the gluteals (gluteus maximus or medius) and infraspinatus on the same side.

Exclusion Criteria:

* neurologic conditions (neuropathy, myopathy)
* use of medication (antidepressants, opioids) and/or acute cervico-thoracic injury (whiplash, facet irritation, acute discopathy) that could directly influence normal somatosensory processing at the C5 segment [Srbely]

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-12; Primary Completion 2023-08 (Actual); Study Completion 2023-08 (Actual)

PRIMARY OUTCOMES:
pressure sensitivity (pain pressure threshold) | 1 week
  Pain pressure threshold values as measured with algometer

SECONDARY OUTCOMES:
Low back pain as measured with visual analog scale (VAS) | 1 week
  a 100 mm line with anchors on the left ('no pain') and on the right ('worst pain imaginable')
modified Oswestry Disability Questionnaire (mOSW) | 1 week
  A 10-item questionnaire assessing low back pain-related disability
15-point Global Rating of Change Scale (GRoC) | 1 week
  A single item questionnaire, where the patient has to quantify his/her improvement or deterioration over time by choosing one of 15 possible answers.

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike H Mitchell, PT, PhD, Principal Investigator — Brigham Young University
Locations (1):
- Brigham Young University Athletics, Provo, Utah, United States

IPD SHARING:
Plan to Share IPD: No
Data will not be shared with any other researcher

REFERENCES:
- [Result] Dunning J, Butts R, Mourad F, Young I, Flannagan S, Perreault T. Dry needling: a literature review with implications for clinical practice guidelines. Phys Ther Rev. 2014 Aug;19(4):252-265. doi: 10.1179/108331913X13844245102034. PMID 25143704
- [Result] Bron C, Dommerholt JD. Etiology of myofascial trigger points. Curr Pain Headache Rep. 2012 Oct;16(5):439-44. doi: 10.1007/s11916-012-0289-4. PMID 22836591
- [Result] Hong CZ, Simons DG. Pathophysiologic and electrophysiologic mechanisms of myofascial trigger points. Arch Phys Med Rehabil. 1998 Jul;79(7):863-72. doi: 10.1016/s0003-9993(98)90371-9. PMID 9685106
- [Result] Shah JP, Gilliams EA. Uncovering the biochemical milieu of myofascial trigger points using in vivo microdialysis: an application of muscle pain concepts to myofascial pain syndrome. J Bodyw Mov Ther. 2008 Oct;12(4):371-384. doi: 10.1016/j.jbmt.2008.06.006. Epub 2008 Aug 13. PMID 19083696
- [Result] Quintner JL, Bove GM, Cohen ML. A critical evaluation of the trigger point phenomenon. Rheumatology (Oxford). 2015 Mar;54(3):392-9. doi: 10.1093/rheumatology/keu471. Epub 2014 Dec 3. PMID 25477053
- [Result] Quintner JL, Cohen ML. Referred pain of peripheral nerve origin: an alternative to the "myofascial pain" construct. Clin J Pain. 1994 Sep;10(3):243-51. doi: 10.1097/00002508-199409000-00012. PMID 7833584
- [Result] Fernandez-de-las-Penas C, Cuadrado ML, Arendt-Nielsen L, Simons DG, Pareja JA. Myofascial trigger points and sensitization: an updated pain model for tension-type headache. Cephalalgia. 2007 May;27(5):383-93. doi: 10.1111/j.1468-2982.2007.01295.x. Epub 2007 Mar 14. PMID 17359516
- [Result] Niddam DM, Chan RC, Lee SH, Yeh TC, Hsieh JC. Central representation of hyperalgesia from myofascial trigger point. Neuroimage. 2008 Feb 1;39(3):1299-306. doi: 10.1016/j.neuroimage.2007.09.051. Epub 2007 Oct 11. PMID 17999939
- [Result] Tough EA, White AR, Cummings TM, Richards SH, Campbell JL. Acupuncture and dry needling in the management of myofascial trigger point pain: a systematic review and meta-analysis of randomised controlled trials. Eur J Pain. 2009 Jan;13(1):3-10. doi: 10.1016/j.ejpain.2008.02.006. Epub 2008 Apr 18. PMID 18395479
- [Result] Tekin L, Akarsu S, Durmus O, Cakar E, Dincer U, Kiralp MZ. The effect of dry needling in the treatment of myofascial pain syndrome: a randomized double-blinded placebo-controlled trial. Clin Rheumatol. 2013 Mar;32(3):309-15. doi: 10.1007/s10067-012-2112-3. Epub 2012 Nov 9. PMID 23138883
- [Result] Kietrys DM, Palombaro KM, Azzaretto E, Hubler R, Schaller B, Schlussel JM, Tucker M. Effectiveness of dry needling for upper-quarter myofascial pain: a systematic review and meta-analysis. J Orthop Sports Phys Ther. 2013 Sep;43(9):620-34. doi: 10.2519/jospt.2013.4668. PMID 23756457
- [Result] Boyles R, Fowler R, Ramsey D, Burrows E. Effectiveness of trigger point dry needling for multiple body regions: a systematic review. J Man Manip Ther. 2015 Dec;23(5):276-93. doi: 10.1179/2042618615Y.0000000014. PMID 26955257
- [Result] Streitberger K, Kleinhenz J. Introducing a placebo needle into acupuncture research. Lancet. 1998 Aug 1;352(9125):364-5. doi: 10.1016/S0140-6736(97)10471-8. PMID 9717924
- [Result] Srbely JZ, Dickey JP, Lee D, Lowerison M. Dry needle stimulation of myofascial trigger points evokes segmental anti-nociceptive effects. J Rehabil Med. 2010 May;42(5):463-8. doi: 10.2340/16501977-0535. PMID 20544158
- [Result] Copay AG, Glassman SD, Subach BR, Berven S, Schuler TC, Carreon LY. Minimum clinically important difference in lumbar spine surgery patients: a choice of methods using the Oswestry Disability Index, Medical Outcomes Study questionnaire Short Form 36, and pain scales. Spine J. 2008 Nov-Dec;8(6):968-74. doi: 10.1016/j.spinee.2007.11.006. Epub 2008 Jan 16. PMID 18201937
- [Result] Kamper SJ, Maher CG, Mackay G. Global rating of change scales: a review of strengths and weaknesses and considerations for design. J Man Manip Ther. 2009;17(3):163-70. doi: 10.1179/jmt.2009.17.3.163. PMID 20046623
- [Result] Chou LW, Hsieh YL, Kuan TS, Hong CZ. Needling therapy for myofascial pain: recommended technique with multiple rapid needle insertion. Biomedicine (Taipei). 2014;4(2):13. doi: 10.7603/s40681-014-0013-2. Epub 2014 Aug 2. PMID 25520926
- [Result] Childs JD, Piva SR, Fritz JM. Responsiveness of the numeric pain rating scale in patients with low back pain. Spine (Phila Pa 1976). 2005 Jun 1;30(11):1331-4. doi: 10.1097/01.brs.0000164099.92112.29. PMID 15928561